CLINICAL TRIAL: NCT01708564
Title: A Phase 1b, Dose Escalation Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Coagulation Factor VIIa (Recombinant) in Congenital Hemophilia A or B Patients
Brief Title: A Phase I Safety, Pharmacokinetics and Pharmacodynamics Study of Recombinant Factor VIIa in Adult Patients With Hemophilia A or B
Acronym: rhFVIIa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: rEVO Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GTC-FVIIa-005-11; 2012-002285-13 (EudraCT Number)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 10 patients administered a single low dose of rhFVIIa
  Interventions: Biological: rhFVIIa
- Cohort 2 (Experimental): 10 patients administered a single intermediate dose of rhFVIIa
  Interventions: Biological: rhFVIIa
- Cohort 3 (Experimental): 10 patients administered a single high dose of rhFVIIa
  Interventions: Biological: rhFVIIa

INTERVENTIONS:
Biological: rhFVIIa — Patients will be administered low, intermediate and high doses of rhFVIIa
  Other Names: Coagulation Factor VIIa (Recombinant)

SUMMARY:
This study will assess the pharmacokinetics and pharmacodynamics of rhFVIIa at three dose levels. The results will help identify the most optimal doses to take forward to the Phase 2/3 studies where bleedings in hemophilia patients with inhibitors will be treated with rhFVIIa.

ELIGIBILITY:
Inclusion Criteria:

1. be male with a diagnosis of moderate or severe congenital hemophilia A and/or B (with or without inhibitors)
2. be 18 years or older, up to and including 75 years of age
3. be capable of understanding and willing to comply with the conditions of the protocol
4. have read, understood and provided written informed consent

Exclusion Criteria:

1. have any coagulation disorder other than hemophilia A or B
2. have a body weight >105 kg (231 lb)
3. be immuno-suppressed (i.e., the patient should not receive systemic immunosuppressive medication <30 days prior to enrollment, CD4 counts at screening should be >200/µl)
4. have a known allergy or hypersensitivity to rabbits
5. have platelet count <100,000/mL
6. have had within one month prior to first administration of the study drug in this study a major surgical procedure (e.g. orthopedic, abdominal)
7. have an active, ongoing bleeding for which the patient is being treated, or treatment for a bleeding was stopped within 24 hours of the time of study drug administration
8. have received a Factor VII or FVIIa containing product (either plasma derived or recombinant) within 72 hours prior to any study drug administration
9. have received an investigational drug within 30 days of the first study drug administration, or is expected to receive such drug during participation in this study
10. have a clinically relevant hepatic (hepatic enzymes >3 times the upper limit of normal) and/or renal impairment (creatinine >2 times the upper limit of normal)
11. have a history of arterial and/or venous thromboembolic events (such as myocardial infarction, ischemic strokes, transient ischemic attacks, deep venous thrombosis or pulmonary embolism) within 2 years prior to first dose of study drug, have an arterial stent in place or have clinically significant atherosclerotic disease (e.g., angina pectoris, peripheral vascular disease)
12. use any anticoagulant for arterial/venous obstructions and/or atrial fibrillation within 7 days prior to first study drug administration
13. have an active malignancy (those with non-melanoma skin cancer are allowed)
14. have any life-threatening disease or other disease or condition which, according to the investigator's judgment, could imply a potential hazard to the patient, interfere with the trial participation or trial outcome

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Factor VIIa concentration in patient plasma as measured by FVIIa PK and PD assays | Up to 36 hours of dosing

SECONDARY OUTCOMES:
Incidence of patients with treatment emergent adverse events | Up to 28 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Johan Frieling, MD,PhD, Study Director — rEVO Biologics
Locations (3):
- United States (2):
  - UC Davis Health System Internal Medicine: Hematology & Oncology, Sacramento, California
  - RUSH Hemophilia & Thrombophilia Center, Chicago, Illinois
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Carcao M, Hermans C, Giermasz A, Kessler C, Miesbach W, Quon D, Windyga J, Mahlangu J. Safety and Use of Eptacog Beta 225 microg/kg in Patients With Haemophilia A or B With Inhibitors. Haemophilia. 2025 Sep;31(5):957-965. doi: 10.1111/hae.70083. Epub 2025 Jul 17. PMID 40674256